CLINICAL TRIAL: NCT06976515
Title: Initial Cohort Study for Remote Investigation of Eye Dryness: A Pilot and Feasibility Study
Brief Title: Study for Remote Investigation of Evaporative Dry Eye Disease
Acronym: I CRIED
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: That Man May See, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 25-43371
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Evaporative Loss Dry Eye Disease
Keywords: Dry Eye; Evaporative Loss Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Self-collected tear production measurement. This is called a Schirmer test. Self-collected eyelid swab. Only the remote recruitment group will be asked to perform this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UCSF Recruitment Group: For this feasibility trial any patient identified in the eye clinics of the UCSF Department of Ophthalmology, Optometry, or Proctor Foundation clinic with evaporative dry eye as a primary diagnosis will be queried with regard to participation interest. Participants are recruited in person but are consented remotely. To mimic a larger, scalable, future-anticipated recruitment strategy, interested participants will be asked to scan a QR code to indicate interest in the study. Study information will be posted in clinic rooms and waiting rooms.
- Remote Recruitment Group: Anterior Segment Delegates of Optometry have specialty training in ocular surface disease and are located across the entire United States. Study information will be sent to Anterior Segment Delegates of the American Board of Optometry who have expressed interest in this study design. Recruitment sheets will be offered for them to post in their clinics and waiting rooms. Once an Anterior Segment delegate has confirmed dry eye disease in the interested participant, they will scan the study QR code to indicate interest in the study.
  Alternatively, if sample size is not met we will recruit through ophthalmology listservs. All participants recruited through anterior segment delegates or listservs will give permission for their eye doctor to be contacted to confirm evaporative dry eye is their primary diagnosis and that no exclusion criteria exist.

SUMMARY:
Dry eye disease is a common problem that can make your eyes feel uncomfortable and affect your vision, making daily tasks harder. Many past studies on dry eye treatments haven't worked well because they didn't include enough people or different types of people. Doing studies at home instead of at the doctor's office can help more people join and make it easier to find out which treatments really work.

DETAILED DESCRIPTION:
This is a feasibility study, this is not an interventional study. This proposal outlines a novel approach to the study of dry eye disease through a decentralized clinical trial design. This non-interventional planning and feasibility proposal shifts the focus of dry eye disease study away from doctors' offices and into participants' home environments. Subjective dry eye disease symptoms are collected remotely, electronically, and sequentially. Self-collected ocular surface samples are collected in two ways: with a self-collected Schirmer strips and with a self-collected ocular surface swab of the eyelid margin and conjunctiva. All study materials are mailed to participants' homes. Self-collected ocular surface samples are placed in study vials and return-mailed by the participant to a central location, UCSF Proctor Foundation laboratory. Here, the samples are processed for RNA-deep sequencing which allows for host transcriptomic analysis. To mimic repeat ocular surface collection after a future dry eye disease intervention, Schirmer strips and ocular surface self-swabbing will be repeated after 4 weeks. This decentralized approach to dry eye disease study promotes patient engagement, recruitment, communication, and participant diversity and also seeks to identify new objective markers of dry eye disease efficacy that can be collected remotely.

ELIGIBILITY:
Inclusion Criteria:

* Evaporative loss dry eye disease will be confirmed by screening clinical examination. Patients with evaporative loss dry eye disease will have minimal to no corneal staining and have normal aqueous (water) tear production. Eligible patients with evaporative loss dry eye disease over the age of 18 will be offered study participation.
* There will be no ethnic restrictions on enrollment. All adults (18 years of age or older) with evaporative loss dry eye disease regardless of race or ethnicity will be recruited for participation.
* All adults (18 years of age or older) with evaporative loss dry eye disease , regardless of sex/gender are eligible for recruitment. Women will not be excluded if they are pregnant or breastfeeding.
* All adults age 18 or older with evaporative loss dry eye disease will be recruited for participation. Dry eye disease is not common in the pediatric population and younger children would require assistance with electronic symptom logging and self-performed ocular surface sample collection. Therefore, this study of feasibility of decentralized dry eye disease study will exclude children.
* No treatment is administered in this non-interventional feasibility trial, therefore if pregnant women have dry eye they can participate with no risk to the fetus.

Exclusion Criteria:

* Patients with keratoconjunctivitis sicca (clinically significant decrease in aqueous production) will not be included. This is because the population with this dry eye disease subtype is at higher risk for corneal epithelial breakdown and ocular surface infection.
* Patients unwilling to measure their own tear production at home will be excluded.
* Patients without internet access or reasonable proximity/access to a post box will be excluded.
* Eyedrop use is not an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study will enroll patients over the age of 18 with evaporative loss dry eye disease with minimal to no corneal staining and normal tear production.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Completion of Surveys and Receipt of Samples | 4 weeks
  The primary outcome is the rate of successful completion of the OSDI and SPEED surveys at two time points and the receipt of two clinical samples from two time points.

SECONDARY OUTCOMES:
Comparison of results of remote symptom surveys over time without intervention to inform variability | 4 weeks
Quantification of Recoverable Human mRNA from Self-Collected Schirmer Strips for Transcriptome Analysis | 4 weeks
  The measurement used to assess this outcome will be the quantity of recoverable human mRNA extracted from self-collected Schirmer strips, expressed as the total number of high-quality, aligned transcript reads per sample after RNA sequencing.
Assessment of Intra-Participant Variability in Inflammatory Cytokine Gene Expression in Tears Over Time Using RNA Sequencing. | 4 weeks
  The measurement will be the expression levels of selected inflammatory cytokine genes, quantified as normalized transcript read counts derived from RNA sequencing data. Gene expression levels will be assessed at two time points, 4 weeks apart, with no intervention. Paired comparisons will be made to evaluate intra-participant variability and overall variance across the cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Gerami Seitzman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] "Uninformative research" is the global health crisis you've never heard of. The Gates Foundation. Accessed September 23, 2024. https://www.gatesfoundation.org/ideas/articles/deworm3-clinical-trialsshow- the-value-of-informed-researchhttps://www.gatesfoundation.org/ideas/articles/deworm3-clinicaltrials- show-the-value-of-informed-research
- [Background] Yu J, Asche CV, Fairchild CJ. The economic burden of dry eye disease in the United States: a decision tree analysis. Cornea. 2011 Apr;30(4):379-87. doi: 10.1097/ICO.0b013e3181f7f363. PMID 21045640
- [Background] Stapleton F, Alves M, Bunya VY, Jalbert I, Lekhanont K, Malet F, Na KS, Schaumberg D, Uchino M, Vehof J, Viso E, Vitale S, Jones L. TFOS DEWS II Epidemiology Report. Ocul Surf. 2017 Jul;15(3):334-365. doi: 10.1016/j.jtos.2017.05.003. Epub 2017 Jul 20. PMID 28736337
- [Background] McCann P, Abraham AG, Mukhopadhyay A, Panagiotopoulou K, Chen H, Rittiphairoj T, Gregory DG, Hauswirth SG, Ifantides C, Qureshi R, Liu SH, Saldanha IJ, Li T. Prevalence and Incidence of Dry Eye and Meibomian Gland Dysfunction in the United States: A Systematic Review and Meta-analysis. JAMA Ophthalmol. 2022 Dec 1;140(12):1181-1192. doi: 10.1001/jamaophthalmol.2022.4394. PMID 36301551
- [Background] Sehrawat O, Noseworthy PA, Siontis KC, Haddad TC, Halamka JD, Liu H. Data-Driven and Technology-Enabled Trial Innovations Toward Decentralization of Clinical Trials: Opportunities and Considerations. Mayo Clin Proc. 2023 Sep;98(9):1404-1421. doi: 10.1016/j.mayocp.2023.02.003. PMID 37661149
- [Background] Hanley DF Jr, Bernard GR, Wilkins CH, Selker HP, Dwyer JP, Dean JM, Benjamin DK Jr, Dunsmore SE, Waddy SP, Wiley KL Jr, Palm ME, Mould WA, Ford DF, Burr JS, Huvane J, Lane K, Poole L, Edwards TL, Kennedy N, Boone LR, Bell J, Serdoz E, Byrne LM, Harris PA. Decentralized clinical trials in the trial innovation network: Value, strategies, and lessons learned. J Clin Transl Sci. 2023 Jul 25;7(1):e170. doi: 10.1017/cts.2023.597. eCollection 2023. PMID 37654775
- [Background] Jean-Louis G, Seixas AA. The value of decentralized clinical trials: Inclusion, accessibility, and innovation. Science. 2024 Aug 23;385(6711):eadq4994. doi: 10.1126/science.adq4994. Epub 2024 Aug 23. PMID 39172847
- [Background] McCann P, Kruoch Z, Lopez S, Malli S, Qureshi R, Li T. Interventions for Dry Eye: An Overview of Systematic Reviews. JAMA Ophthalmol. 2024 Jan 1;142(1):58-74. doi: 10.1001/jamaophthalmol.2023.5751. PMID 38127364